CLINICAL TRIAL: NCT00538486
Title: Which is the Best Treatment for Non-diabetic Hypertension With Obesity: Telmisartan, Amlodipine or Candesartan, Alone or Plus MEtformin? (HOT-ACME 1)
Brief Title: A Randomized, Double-Blind, Active Control Trial Comparing Effects of Telmisartan, Candesartan and Amlodipine, Alone or Plus Metformin, on Non-Diabetic, Obese Hypertensive Patients
Acronym: HOT-ACME
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Zhiming Zhu, Director of Dept. of Hypertension & Endocrinology, Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HOT-ACME 1
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Hypertension; Obesity
Keywords: Hypertension; Abdominal obesity; Treatment
MeSH Terms: conditions — Hypertension; Obesity; Obesity, Abdominal | interventions — Telmisartan; Metformin; candesartan; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Group T (Experimental): Telmisartan
  Interventions: Drug: Telmisartan
- Group T+M (Experimental): Telmisartan plus Metformin
  Interventions: Drug: Telmisartan plus Metformin
- Group C (Experimental): Candesartan
  Interventions: Drug: Candesartan
- Group C+M (Experimental): Candesartan pus Metformin
  Interventions: Drug: Candesartan plus Metformin
- Group A (Active Comparator): Amlodipine
  Interventions: Drug: Amlodipine
- Group A+M (Experimental): Amlodipine plus Metformin
  Interventions: Drug: Amlodipine plus Metformin

INTERVENTIONS:
Drug: Telmisartan plus Metformin — Telmisartan 80mg 1/d, Metformin 250mg 2/d
  Arms: Group T+M
Drug: Telmisartan — Telmisartan 80mg 1/d
  Other Names: Telmisartan Alone
  Arms: Group T
Drug: Candesartan — Candesartan 8mg daily
  Other Names: Candesartan Alone
  Arms: Group C
Drug: Candesartan plus Metformin — Candesartan 8mg 1/d Metformin 250mg 2/d
  Arms: Group C+M
Drug: Amlodipine — Amlodipine 5mg 1/d
  Other Names: Amlodipine alone
  Arms: Group A
Drug: Amlodipine plus Metformin — Amlodipine 5mg 1/d, Metformin 250mg 2/d
  Arms: Group A+M

SUMMARY:
The epidemic of obesity is associated with a considerable rise in the incidence of the metabolic syndrome, type 2 diabetes mellitus, and hypertension. Insulin resistance plays an important role in the pathogenesis of obesity related hypertension. These patients are at high risk to suffer from cardiovascular events. However, current guidelines for treatment of hypertension do not provide specific recommendation for the pharmacotherapy of obese hypertensive patients due to lack of prospective randomized intervention studies in non-diabetic obese hypertensive patients.

Aside from their antihypertensive effects, angiotensin II receptor blockers (ARB) were shown to improve insulin sensitivity. Furthermore, metformin is commonly used to treat the obese type 2 diabetes mellitus. Metformin can also lower body weight and increase insulin sensitivity. In a prospective, double-blind, double-dummy, randomized, parallel-group study, we will evaluate the effects of ARB (telmisartan and candesartan) or amlodipine combination with metformin on weight gain, visceral fat, and metabolic parameters in obese hypertensive patients without diabetes mellitus compared with obese hypertensives on ARB or amlodipine treatment alone. This study will help to develop future comprehensive treatment strategies and guidelines for obesity related hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Grade 1 or 2 hypertension: 140mmHg≤SBP<180mmHg, and/or 90mmHg≤DBP<110mmHg
* Waist circumference higher than 90cm in men, 80cm in women

Exclusion Criteria:

* Diabetes
* Grade 3 hypertension: SBP≥180mmHg, or DBP≥110mmHg
* known allergy or hypersensitivity to trial drugs
* Myocardial infarction or cerebrovascular accident in the year preceding the trial
* Clinical Congestive Heart Failure
* History of hepatitis or cirrhosis
* History of kidney disease

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2008-02; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | Baseline, 24 weeks(End of trial)
Metabolic profiles, including lipid profile and blood glucose | Baseline, 24 weeks(End of trial)

SECONDARY OUTCOMES:
Abdominal fat assessed by CT | Baseline, 24 weeks(End of trial)
Obesity parameters, including waist circumference (WC) and body mass index (BMI) | Baseline, 24 weeks(End of trial)
Insulin resistance assessed by fasting serum insulin and HOMA-IR | Baseline, 24 weeks(End of trial)
Incidents of side effects between groups | Baseline, 24 weeks(End of trial)

CONTACTS AND LOCATIONS:
Overall Officials: Zhiming Zhu, MD, PhD, Principal Investigator — The third hospital affiliated to the Third Military Medical University. China; Zhiming Zhu, MD, PhD, Study Director — The third hospital affiliated to the Third Military Medical University. China
Locations (1):
- The third hospital affiliated to the Third Military Medical University, Chongqing, China

REFERENCES:
- [Result] He H, Zhao Z, Chen J, Ni Y, Zhong J, Yan Z, Li Y, Liu D, Pletcher MJ, Zhu Z. Metformin-based treatment for obesity-related hypertension: a randomized, double-blind, placebo-controlled trial. J Hypertens. 2012 Jul;30(7):1430-9. doi: 10.1097/HJH.0b013e328353e249. PMID 22525206